CLINICAL TRIAL: NCT04199351
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 171 in Subjects With Obesity
Brief Title: Single and Multiple Ascending Dose Study of AMG 171 in Subjects With Obesity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen determined the totality of the data does not support continuation of AMG 171 development program for treatment of Obesity. No safety concerns identified.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20180224
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): AMG 171 or placebo, 2 SAD cohorts
  Interventions: Drug: AMG 171; Drug: Placebo
- Part B (Experimental): AMG 171 or placebo, 1 MAD cohort
  Interventions: Drug: AMG 171; Drug: Placebo
- Part C (Experimental): AMG 171 or placebo, 3 titration cohorts
  Interventions: Drug: AMG 171; Drug: Placebo

INTERVENTIONS:
Drug: AMG 171 — 2 SAD cohorts of 8 subjects per cohort randomized 3:1 in Part A; 1 cohort of 8 subjects 3:1 ratio in Part B; and 24 subjects enrolled into 1 of 3 cohorts with 8 subjects randomized to receive 2 to 3 consecutive doses (titration) 3:1 ratio in Part C.
Drug: Placebo — AMG 171 placebo

SUMMARY:
To assess the safety and tolerability of AMG 171 as single or multiple doses in subjects with obesity

ELIGIBILITY:
Inclusion Criteria

* Males and females with ages between 18 and 65 years old, inclusive
* Except for obesity, otherwise healthy
* Body mass index (BMI) greater than or equal to 30.0 kg/m2 and less than or equal to 40.0 kg/m2 at screening
* Other Inclusion criteria may apply

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study
* Women of childbearing potential
* History or evidence of a clinically significant disorder, condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Other Exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, LLC, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a datasharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 study centers in the United States, and participated from 13 December 2019 to 10 September 2021.
Pre-assignment Details: Participants were enrolled into single ascending dose (SAD) cohorts in Part A (Cohorts 1 and 1b), a multiple dosing cohort in Part B (Cohort 2), and step dosing cohorts in Part C (Cohorts 3 - 5). Three doses were given: Dose A (low dose), Dose B (intermediate dose), and Dose C (high dose).
Groups:
- Placebo (Cohorts 1 and 1b): Participants in Part A Cohorts 1 and 1b were randomized to receive a single subcutaneous (SC) dose of placebo on Day 1.
- Cohort 1 (Part A): AMG 171 Dose A: Participants were randomized to receive AMG 171 Dose A as a single SC dose on Day 1.
- Cohort 1b (Part A): AMG 171 Dose B: Participants were randomized to receive AMG 171 Dose B as a single SC dose on Day 1.
- Placebo (Cohort 4 Replaced): Participants enrolled in Part C Cohort 4 received compromised or expired investigational product (IP). These participants were randomized to receive placebo on Day 1, Day 15, and on Day 29, as SC doses.
- Placebo (Cohorts 2-5): Participants in Parts B and C (Cohorts 2-5) were randomized to receive multiple SC doses of placebo.
- Cohort 2 (Part B): AMG 171 Dose A Q2W: Participants were randomized to receive AMG 171 Dose A every 2 weeks (Q2W) on Days 1, 15, 29, 43, 57, and 71, as SC doses.
- Cohort 3 (Part C): AMG 171 Dose A/Dose B: Participants were randomized to receive AMG 171 Dose A on Day 1 and Dose B on Day 15, as SC doses.
- Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C: Participants were randomized to receive AMG 171 Dose A on Day 1, Dose B on Day 15, and Dose C on Day 29, as SC doses.
- Cohort 5 (Part C): AMG 171 Dose A/Dose B: Participants were randomized to receive AMG 171 Dose A on Day 1 and Dose B on Day 8, as SC doses.
- Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C: Participants enrolled in Part C Cohort 4 received compromised or expired IP. These participants were randomized to receive AMG 171 Dose A on Day 1, Dose B on Day 15, and Dose C on Day 29, as SC doses.
Period: Overall Study
Arm/Group | Placebo (Cohorts 1 and 1b) | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B | Placebo (Cohort 4 Replaced) | Placebo (Cohorts 2-5) | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C
Started | 4 | 7 | 6 | 2 | 8 | 7 | 8 | 6 | 6 | 6
Completed | 4 | 6 | 5 | 0 | 7 | 2 | 6 | 6 | 3 | 0
Not Completed | 0 | 1 | 1 | 2 | 1 | 5 | 2 | 0 | 3 | 6
Not completed — Decision by sponsor | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 4 | 2 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Cohort 1 and 1b): Participants in Part A Cohorts 1 and 1b were randomized to receive a single SC dose of placebo on Day 1.
- Placebo (Cohort 4 Replaced): Participants enrolled in Part C Cohort 4 received compromised or expired IP. These participants were randomized to receive placebo on Day 1, Day 15, and on Day 29, as SC doses.
- Cohort 2 (Part B): AMG 171 Dose A Q2W: Participants were randomized to receive AMG 171 Dose A Q2W on Days 1, 15, 29, 43, 57, and 71, as SC doses.
- Total: Total of all reporting groups
Arm/Group | Placebo (Cohort 1 and 1b) | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B | Placebo (Cohort 4 Replaced) | Placebo (Cohorts 2-5) | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C | Total
Number analyzed (Participants) | 4 | 7 | 6 | 2 | 8 | 7 | 8 | 6 | 6 | 6 | 60
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 64 years | 4 | 7 | 6 | 2 | 8 | 7 | 8 | 6 | 6 | 6 | 60
  ≥ 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 3 | 2 | 16
  Male | 2 | 7 | 5 | 1 | 6 | 5 | 6 | 5 | 3 | 4 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 2 | 4 | 3 | 2 | 6 | 1 | 6 | 34
  Not Hispanic or Latino | 1 | 3 | 3 | 0 | 4 | 4 | 6 | 0 | 5 | 0 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 1 | 2 | 0 | 4 | 4 | 3 | 0 | 4 | 3 | 21
  White | 4 | 6 | 4 | 2 | 3 | 3 | 5 | 6 | 2 | 3 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with study treatment. A serious AE (SAE) was an AE meeting at least 1 of the following serious criteria: fatal, life-threatening, required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability; congenital anomaly/birth defect; other medically important serious event. Clinically significant changes from baseline in laboratory safety tests, vital sign assessments, and 12-lead electrocardiogram assessments were included as TEAEs.
Time Frame: From first dose of IP to end of study, up to Day 207
Population: The safety analysis set included all participants who received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Cohort 1 and 1b) | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B | Placebo (Cohort 4 Replaced) | Placebo (Cohorts 2-5) | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C
Number analyzed (Participants) | 4 | 7 | 6 | 2 | 8 | 7 | 8 | 6 | 6 | 6
Participants
  Any TEAEs | 0 | 5 | 6 | 0 | 3 | 7 | 5 | 5 | 5 | 5
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to IP discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for AMG 171: SAD Cohorts 1 and 1b
Description: Serum concentrations of AMG 171 were determined using a validated assay. Noncompartmental analysis was performed for estimation of pharmacokinetic (PK) parameters. Concentrations below the lower limit of quantification (LLOQ) (50.0 ng/mL) were set to zero before data analysis.
Time Frame: Cohorts 1 and 1b: pre-dose Day 1; 1, 2, 4, and 8 hours post-dose Day 1, Days 2 up to Day 120
Population: The PK analysis set included all participants who received at least 1 dose of AMG 171 for whom at least 1 PK parameter could be adequately estimated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B
Number analyzed (Participants) | 7 | 6
ng/mL | 697 (405) | 1740 (759)

3. Secondary Outcome: Cmax for AMG 171: MAD Cohorts 2 - 5
Description: Serum concentrations of AMG 171 were determined using a validated assay. Noncompartmental analysis was performed for estimation of PK parameters. Concentrations below the LLOQ (50.0 ng/mL) were set to zero before data analysis.
Time Frame: Cohort 2: pre-dose Days 1, 15, 29, 43, 57, 71; post-dose Days 5 up to 207; Cohort 3: pre-dose Days 1, 15; post-dose Days 2 up to 85; Cohort 4: pre-dose Days 1, 15, 29; post-dose Days 2 up to 113; Cohort 5: pre-dose Days 1, 8; post-dose Days 2 up to 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B
Number analyzed (Participants) | 7 | 8 | 6 | 6
ng/mL
  Day 1 | 695 (229) | 847 (522) | 455 (335) | 769 (470)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 4
  Day 8 |  |  |  | 2550 (1820)
  Day 15: number analyzed (Participants) | 0 | 6 | 6 | 0
  Day 15 |  | 1350 (670) | 1760 (1080) |
  Day 29: number analyzed (Participants) | 0 | 0 | 6 | 0
  Day 29 |  |  | 3960 (1600) |
  Day 71: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 71 | 1490 (702) |  |  |

4. Secondary Outcome: Time of Cmax (Tmax) for AMG 171: SAD Cohorts 1 and 1b
Description: as for outcome 3
Time Frame: Cohorts 1 and 1b: pre-dose Day 1; 1, 2, 4, and 8 hours post-dose Day 1, Days 2 up to Day 120
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B
Number analyzed (Participants) | 7 | 6
hours | 120 [47 to 120] | 120 [72 to 120]

5. Secondary Outcome: Tmax for AMG 171: MAD Cohorts 2 - 5
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B
Number analyzed (Participants) | 7 | 8 | 6 | 6
hours
  Day 1 | 93 [91 to 310] | 60 [19 to 310] | 84 [48 to 190] | 58 [21 to 160]
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 4
  Day 8 |  |  |  | 82 [45 to 220]
  Day 15: number analyzed (Participants) | 0 | 6 | 6 | 0
  Day 15 |  | 72 [48 to 310] | 96 [48 to 120] |
  Day 29: number analyzed (Participants) | 0 | 0 | 6 | 0
  Day 29 |  |  | 110 [72 to 120] |
  Day 71: number analyzed (Participants) | 3 | 0 | 0 | 0
  Day 71 | 72 [61 to 73] |  |  |

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Infinity (AUCinf) for AMG 171: SAD Cohorts 1 and 1b
Description: as for outcome 3
Time Frame: Cohorts 1 and 1b: pre-dose Day 1; 1, 2, 4, and 8 hours post-dose Day 1, Days 2 up to Day 120
Population: The PK analysis set included all participants who received at least 1 dose of AMG 171 for whom at least 1 PK parameter could be adequately estimated. Participants with available data are included.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B
Number analyzed (Participants) | 6 | 5
hours*ng/mL | 285000 (72200) | 792000 (324000)

7. Secondary Outcome: AUC From Time 0 to 14 Days (AUC0-14) for AMG 171: MAD Cohorts 2 - 4
Description: as for outcome 3
Time Frame: Cohort 2: pre-dose Days 1, 15, 29, 43, 57, 71; post-dose Days 5 up to 207; Cohort 3: pre-dose Days 1, 15; post-dose Days 2 up to 85; Cohort 4: pre-dose Days 1, 15, 29; post-dose Days 2 up to 113
Population: The PK analysis set included all participants who received at least 1 dose of AMG 171 for whom at least 1 PK parameter could be adequately estimated. Participants with data available are included.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C
Number analyzed (Participants) | 3 | 7 | 6
hours*ng/mL
  Day 1: number analyzed (Participants) | 3 | 7 | 5
  Day 1 | 201000 (36400) | 205000 (123000) | 133000 (74000)
  Day 8: number analyzed (Participants) | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 0 | 6 | 6
  Day 15 |  | 362000 (160000) | 440000 (261000)
  Day 29: number analyzed (Participants) | 0 | 0 | 6
  Day 29 |  |  | 1050000 (429000)
  Day 71: number analyzed (Participants) | 3 | 0 | 0
  Day 71 | 375000 (120000) |  |

8. Secondary Outcome: AUC From Time 0 to 7 Days (AUC0-7) for AMG 171: MAD Cohort 5
Description: as for outcome 3
Time Frame: Cohort 5: pre-dose Days 1, 8; post-dose Days 2 up to 85
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Cohort 5 (Part C): AMG 171 Dose A/Dose B
Number analyzed (Participants) | 4
hours*ng/mL
  Day 1: number analyzed (Participants) | 3
  Day 1 | 138000 (47200)
  Day 8 | 351000 (272000)

9. Secondary Outcome: Number of Participants With Anti-AMG 171 Antibodies
Description: Serum samples were tested for binding and neutralizing antibodies against human Growth Differentiation Factor 15. Participants with transiently positive for binding or neutralizing antibodies had a negative result at the participant's last time point tested.
  bAb = binding antibody; nAb = neutralizing antibody; +ve = positive; -ve = negative; BL = baseline.
Time Frame: Cohorts 1 and 1b: Day 1 pre-dose, Days 15, 29, 120; Cohort 2: Days 1, 29, 57 pre-dose, Days 15, 85, 207; Cohort 3: Days 1, 15 pre-dose, Days 29, 57, 85; Cohort 4: Days 1, 15, 29 pre-dose, Days 43, 85, 113; Cohort 5: Days 1, 8 pre-dose, Days 29, 57, 85
Population: The safety analysis set included all participants who received at least 1 dose of IP. Data for participants with an on-study result are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Cohort 1 and 1b) | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B | Placebo (Cohort 4 Replaced) | Placebo (Cohorts 2-5) | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C
Number analyzed (Participants) | 2 | 7 | 6 | 0 | 0 | 7 | 8 | 6 | 6 | 0
Participants
  bAb +ve at/before BL | 1 | 1 | 0 |  |  | 0 | 0 | 0 | 0 |
  nAb +ve at/before BL | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 |
  bAb +ve post-BL with -ve/no result at BL | 0 | 1 | 2 |  |  | 1 | 0 | 0 | 1 |
  Transient bAb +ve post-BL with -ve/no result at BL | 0 | 1 | 0 |  |  | 1 | 0 | 0 | 1 |
  nAb +ve post-BL with -ve/no result at BL | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 |
  Transient nAb +ve post-BL with -ve/no result at BL | 0 | 0 | 0 |  |  | 0 | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from informed consent to end of study, up to approximately 235 days. SAEs and other AEs were collected from first dose of IP to end of study, up to Day 207.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. SAEs and other AEs are reported for all participants who received at least one dose of study drug.
Arm/Group | Placebo (Cohort 1 and 1b) | Cohort 1 (Part A): AMG 171 Dose A | Cohort 1b (Part A): AMG 171 Dose B | Placebo (Cohort 4 Replaced) | Placebo (Cohorts 2-5) | Cohort 2 (Part B): AMG 171 Dose A Q2W | Cohort 3 (Part C): AMG 171 Dose A/Dose B | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C | Cohort 5 (Part C): AMG 171 Dose A/Dose B | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7 | 0/6 | 0/2 | 0/8 | 0/7 | 0/8 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7 | 0/6 | 0/2 | 0/8 | 0/7 | 0/8 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 5/7 | 6/6 | 0/2 | 3/8 | 7/7 | 5/8 | 5/6 | 5/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Cohort 1 and 1b) (N=4) | Cohort 1 (Part A): AMG 171 Dose A (N=7) | Cohort 1b (Part A): AMG 171 Dose B (N=6) | Placebo (Cohort 4 Replaced) (N=2) | Placebo (Cohorts 2-5) (N=8) | Cohort 2 (Part B): AMG 171 Dose A Q2W (N=7) | Cohort 3 (Part C): AMG 171 Dose A/Dose B (N=8) | Cohort 4 (Part C): AMG 171 Dose A/Dose B/Dose C (N=6) | Cohort 5 (Part C): AMG 171 Dose A/Dose B (N=6) | Cohort 4 Replaced (Part C): AMG 171 Dose A/Dose B/Dose C (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 6 | 0 | 1 | 5 | 4 | 5 | 4 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 4 | 1 | 2 | 4 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT04199351/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT04199351/SAP_001.pdf